CLINICAL TRIAL: NCT03229083
Title: Monitoring of Treatment Related Toxicities from Oral Targeted Agents and Immunotherapy Among Patients with Advanced Renal Cell Carcinoma (RCC) Using Carevive Software, a Single-Arm Phase II Feasibility Study
Brief Title: Software Monitoring of Treatment Related Toxicities in Advanced Renal Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Chunkit Fung, Doctor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UGUK 17036; UG1CA189961 (NIH)
Record Dates: First submitted 2017-07-18; First posted 2017-07-25 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Advanced Renal Cell Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Use of Carevive software (Experimental): Reporting and management of side effects from oral targeted therapy or immunotherapy, through Carevive software, in patients who have advanced Renal Cell Carcinoma (RCC).
  Interventions: Other: Carevive software

INTERVENTIONS:
Other: Carevive software — In this study, Carevive will deliver a link to subjects so that an online survey can be completed. The survey will occur weekly for the first 12 weeks of the study and will be spaced out to every other week thereafter. The questions will mostly focus on side effects from their cancer therapy, as well as a few questions about drug compliance and healthcare utilization. After completion of the survey, the subject will be given a care plan with at home self-management options for drug-related toxicities.

SUMMARY:
To determine if Carevive software, which monitors treatment-related toxicities and then generates self-care management plans for these symptoms, will be feasible to implement among patients with metastatic renal cell carcinoma (RCC). Additionally for collection of preliminary data on treatment-related toxicities, quality of life, distress level, and drug adherence.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of histologically confirmed renal cell carcinoma of any subtype with either pathological or radiographic evidence of metastatic disease
* Greater than 18 years of age
* A participating Wilmot Cancer Center oncologist has determined that candidate should be started on either oral targeted therapy or immunotherapy for treatment of their advanced RCC; this can be for first-line or any subsequent line therapy
* Able to provide written informed consent
* Proficient in the English language and self-reports as literate
* Must have an active email address or access to a smart device on which text messages can be received

Exclusion Criteria:

* Women cannot be breast-feeding
* Does not have regular access to the internet
* Unable to come to the Wilmot Cancer Center for appointments every 3-4 months for routine visits with their primary oncologist
* Subjects who were on the study previously will not be allowed to re-enroll in the event of a treatment change

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Carevive Survey Usage Rates | 48 weeks
  Carevive software will track subject compliance with survey logins and whether they access the generated care plans. The percentage of times logged in out of the number of study recommended logins will be tabulated. Also, the percentage of times a careplan was accessed out of the number of times it was offered will be determined.
  * To determine the practicality of the intervention, by analyzing the reasons why subjects fail to self-report treatment-related toxicities or utilize software generated care plans after enrollment.
  * To assess the acceptability of this intervention with validated patient reported usability scores of the software.
  * To determine potential implementation obstacles of the intervention, by assessing the reasons eligible study candidates decline participation.
Reasons Participants Do Not Complete Survey or Utilize Care Plans | 48 weeks
  After missing a survey, subjects will be asked the reason at their following login. The reason provided will be sorted into pre-specified categories and presented as a percentage.
Average Usability Score Using the Software Usability Scoring System | 48 weeks
  At the 48 week time point or at the point of subject withdrawal from study, they will be asked to take the System Usability Scale. The survey provides us with a score of between 0 and 40 which is then multiplied by 2.5 to convert to a scale of 0 to 100. A SUS score above a 68 would be considered above average and anything below 68 is below average.
Reasons for Declining Study Participation | 48 weeks
  If a subject declines to participation in the study, he/she will be asked to provide a reason for declination. If willing, we will have them sign a separate consent with a space to write in their reason. The reason provided will be sorted into pre-specified categories and presented as a percentage.

SECONDARY OUTCOMES:
Patient Reported Toxicities Using PRO-CTCAE Questions | 48 weeks
  Patient reported toxicity data will be collected via Carevive surveys weekly for the first 12 weeks and then every other week for another 36 weeks. We will not deliver the PRO-CTCAE in its entirety but will specifically ask about the following common toxicities that are experienced with oral targeted therapy and immunotherapy: diarrhea, nausea, vomiting, fatigue, hand/foot syndrome, rash, abdominal pain, anorexia, mouth sores, cough and shortness of breath.
Clinician Reported Toxicities Using CTCAE | 48 weeks
  Toxicities will also be formally assessed in-office every 3-4 months using CTCAE scoring. The categories chosen are common toxicities that occur with oral targeted therapy and immunotherapy: diarrhea, nausea, vomiting, fatigue, hand/foot syndrome, rash, abdominal pain, appetite, mouth sores, cough and shortness of breath
Quality of Life Determination Using the FKSI-DRS Survey | 48 weeks
  Subjects will be asked to fill out the Functional Assessment of Cancer Therapy-Kidney Symptom Index (FKSI-DRS) at baseline and approximately every 3 months in-office.
Distress Level Using the NCCN Distress Thermometer | 48 weeks
  The subject will be asked to rate their distress level in-office using the NCCN Distress Thermometer, which is a 1 to 10 numerical scale. This will be delivered during routine office visits approximately every 3 months on a tablet.
• Health Care Utilization Assessment By Quantification of Health Care Visits or Hospitalizations | 48 weeks
  Health care utilization will be self-reported by the subject through CareVive software monthly, in addition at the end of the study or at time of withdrawal, a search of the electronic medical record will be performed to determine the number of calls made to oncology care providers and the number of visits to the oncologist during the study period.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester - Wilmot Cancer Institute, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No